CLINICAL TRIAL: NCT01075048
Title: A Randomized, Placebo-Controlled, Phase 1/2 Study Of ARQ 197 in Combination With Irinotecan and Cetuximab in Subjects With Metastatic Colorectal Cancer With Wild-type KRAS Who Have Received Front-Line Systemic Therapy
Brief Title: ARQ 197 in Combination With Chemotherapy in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARQ197-A-U252
Record Dates: First submitted 2010-02-17; First posted 2010-02-24 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer; wild-type KRAS; irinotecan; cetuximab; second-line therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — ARQ 197; Cetuximab; Irinotecan

STUDY DESIGN:
Intervention Model Description: Phase 1 is single group open label with one arm. Phase 2 is parallel, double-blind design with two arms.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 2: Tivantinib, cetuximab, irinotecan (Experimental): Tivantinib in combination with irinotecan and cetuximab.
  Interventions: Drug: Tivantinib; Drug: Cetuximab; Drug: Irinotecan
- Phase 2: Placebo, cetuximab, irinotecan (Placebo Comparator): Placebo in combination with irinotecan and cetuximab
  Interventions: Drug: Placebo; Drug: Cetuximab; Drug: Irinotecan
- Phase 1: Tivantinib, cetuximab, irinotecan (Experimental): Tivantinib in combination with irinotecan and cetuximab.
  Interventions: Drug: Tivantinib; Drug: Cetuximab; Drug: Irinotecan

INTERVENTIONS:
Drug: Tivantinib — ARQ 197 is supplied as a 120-mg capsule, administered twice daily at the dose determined in the Phase 1 portion of the study. Administered until disease progression, unacceptable toxicity or other discontinuation criteria is met.
  Other Names: ARQ 197
  Arms: Phase 1: Tivantinib, cetuximab, irinotecan; Phase 2: Tivantinib, cetuximab, irinotecan
Drug: Placebo — Placebo to match ARQ 197, administered twice daily. Administered until disease progression, unacceptable toxicity or other discontinuation criteria is met.
  Arms: Phase 2: Placebo, cetuximab, irinotecan
Drug: Cetuximab — Cetuximab 500 mg/ m^2 intravenous infusion over 120 minutes at the first cycle, then over 60-minutes at subsequent cycles. Administered on Day 1 and Day 15 of each 28 day cycle. Administered until disease progression, unacceptable toxicity or other discontinuation criteria is met.
Drug: Irinotecan — 60 minutes after cetuximab, Irinotecan 180 mg/m^2 intravenous infusion over 30 - 90 minutes. Administered on Day 1 and Day 15 of each 28 day cycle. Administered until disease progression, unacceptable toxicity or other discontinuation criteria is met.

SUMMARY:
ARQ 197 or placebo in combination with irinotecan and cetuximab in participants with metastatic colorectal cancer (CRC), in participants with wild-type KRAS alleles who have failed front-line systemic therapy, to evaluate the safety, tolerability, and efficacy of ARQ 197, define the recommended dose for Phase 2.

After the recommended dose is determined for Phase 2, participants receive study drug or placebo with irinotecan and cetuximab.

DETAILED DESCRIPTION:
Phase 1/2 Multicenter study:

* Phase 1 portion is open-label to evaluate the safety of ARQ 197 administered in combination with irinotecan and cetuximab.
* Phase 2 portion is designed as a randomized, double-blind placebo-controlled study to assess the efficacy and safety of ARQ 197 or matching placebo administered in combination with irinotecan and cetuximab.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with surgically unresectable locally advanced or metastatic disease who have received one prior line of chemotherapy. (The Phase 1 portion of the study will be open for enrollment for subjects who received 1 or more prior therapies). Both relapsed and refractory CRC are allowed.
2. All participants must express the wild-type form of the gene KRAS.
3. Measurable disease according to RECIST (Response Evaluation Criteria In Solid Tumors) criteria, Version 1.1.
4. Male or female >= to 18 years of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Resolution of any toxic effects of prior therapy (except alopecia) to NCI CTCAE, Version 4.0, grade <= to 1.
7. Adequate bone marrow, liver, and renal functions, defined as:

   * Hemoglobin >= to 9.0 g/dL (transfusion and/or growth factor support allowed).
   * Absolute neutrophil count (ANC) >= to 1.5 x 10^9/L.
   * Platelet count >= to 75 x 10^9/L.
   * Serum creatinine <= to 1.5 x upper limit of normal (ULN) or creatinine clearance >= to 60 mL/min.
   * Alanine transaminase (ALT), aspartate transaminase (AST), and alkaline phosphatase <= to 2.5 x ULN in subjects with no liver metastasis and <= to 5.0 x ULN in participants with liver metastasis.
   * Total bilirubin <= to 1.5 x ULN (<= to 4 x ULN and direct bilirubin <= to 1.5 x ULN is acceptable for subjects with Gilbert's syndrome).
8. Male and female participants of child-bearing potential must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after last investigational drug dose received.
9. All female participants of childbearing potential must each have a negative pregnancy test (serum or urine) result before initiating study treatment.
10. Participants must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an Independent Ethics Committee (IEC) or Institutional Review Board (IRB)-approved informed consent form (ICF) (including HIPAA authorization, if applicable) before performance of any study specific procedures or tests.

Exclusion Criteria:

1. Prior therapy with an Epidermal Growth Factor Receptor (EGFR) inhibitor.
2. History of malignancy other than CRC, unless there is an exception that the malignancy has been cured and no tumor-specific treatment for the malignancy has been administered within the 5 years prior to initiation of study treatment (participants with a history of basal cell carcinoma or benign tumor of cervix can be enrolled if diagnosis and treatment occurred less than 3 years prior to randomization).
3. Anticipation of need for a major surgical procedure or radiation therapy (RT) during the study.
4. Treatment with chemotherapy, radiotherapy, surgery, immunotherapy, biological therapy, or any other investigational anticancer agent within 4 weeks prior to start of study treatment.
5. History of cardiac disease:

   * Congestive heart failure defined as Class II to IV per New York Heart Association (NYHA) classification.
   * Active coronary artery disease (CAD).
   * Previously diagnosed bradycardia or other cardiac arrhythmia defined as Grade 2 or higher according to NCI CTCAE, version 4.0, or uncontrolled hypertension.
   * Myocardial infarction that occurred within 6 months prior to start of study treatment (myocardial infarction that occurred greater than 6 months before the start of study treatment is permitted).
6. Malabsorption syndrome, chronic diarrhea (lasting greater than 4 weeks), inflammatory bowel disease, or partial bowel obstruction.
7. Known metastatic brain or meningeal tumors, unless the participant is greater than 6 months from definitive therapy, has a negative imaging study within 4 weeks of first dose of study treatment, and is clinically stable (no concomitant therapy, including supportive therapy with steroids or anticonvulsant medications) with respect to the tumor at the time of first dose of study treatment.
8. Uncontrolled seizure disorder, spinal cord compression, or carcinomatous meningitis.
9. Pericardial or pleural effusion (eg, requiring drainage) or pericardial involvement with the tumor. Participants with minimal pleural effusion may be eligible upon request by Investigator and approval by Sponsor.
10. Clinically significant active infection that requires antibiotic therapy.
11. Previous administration of ARQ 197.
12. Substance abuse or medical, psychological or social conditions that may, in the opinion of the Investigator, interfere with the participant's participation in the clinical trial or evaluation of the clinical trial results.
13. Any condition that is unstable or that could jeopardize the safety of the subject and the participant's protocol compliance including known human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection.
14. Inability to swallow oral medications.
15. Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2010-01-26 (Actual); Primary Completion 2012-10-12 (Actual); Study Completion 2015-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (40):
- United States (24):
  - Beverly Hills, California
  - Encinitas, California
  - Fountain Valley, California
  - Riverside, California
  - Fort Collins, Colorado
  - Norwich, Connecticut
  - Boynton Beach, Florida
  - Fort Myers, Florida
  - Orlando, Florida
  - Centralia, Illinois
  - Metairie, Louisiana
  - Baltimore, Maryland
  - Hagerstown, Maryland
  - Omaha, Nebraska
  - Buffalo, New York
  - Lake Success, New York
  - Canton, Ohio
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - Seattle, Washington
- France (3):
  - Bayonne
  - Lille
  - Marseille
- Germany (4):
  - Halle
  - Leer
  - Mannheim
  - München
- Italy (3):
  - Milan
  - Reggio Emilia
  - Treviglio
- Russia (6):
  - Chelyabinsk
  - Kursk
  - Moscow
  - Pyatigorsk
  - Saint Petersburg
  - Samara

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 131 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 40 clinic sites (24 in the United States and 16 in Europe).
Pre-assignment Details: Of the 131, 9 participants enrolled into the Phase 1 cohort and 122 participants randomly assigned to ARQ 197 or placebo treatment in Phase 2. In Phase 2, 1 enrolled participant was not treated and therefore not included in the Safety Analysis Set.
Groups:
- Phase 1: ARQ 197+Cetuximab+Irinotecan: Participants received an oral dose of ARQ197 capsules twice daily (BID) with a meal, in escalating doses of 120 milligram (mg), 240 mg, and 360 mg to 3 separate cohorts on Day 1 of Cycle 1 and Cycle 2. Cetuximab 500 mg/m^2 intravenous infusion over 120 minutes at the first cycle, then over 60-minutes at subsequent cycles followed by 60 minutes with irinotecan 180 mg/m^2 intravenous infusion over 30 - 90 minutes. Cetuximab and irinotecan are administered on Day 1 and Day 15 of each 28 day cycle.
- Phase 2: Placebo+Cetuximab+Irinotecan: Participants received placebo twice daily (BID) with cetuximab and irinotecan until disease progression, unacceptable toxicity or other discontinuation. Cetuximab 500 mg/ m^2 intravenous infusion over 120 minutes, then over 60 minutes at subsequent cycles followed 60 minutes later with irinotecan 180 mg/m^2 intravenous infusion over 30 - 90 minutes. Cetuximab and irinotecan are administered on Day 1 and Day 15 of each 28 day cycle.
- Phase 2: ARQ 197+Cetuximab+Irinotecan: Participants received ARQ197 (recommended Phase 2 dose of 720 mg) daily with cetuximab and irinotecan until disease progression, unacceptable toxicity or other discontinuation. Cetuximab 500 mg/m^2 intravenous infusion over 120 minutes at the first cycle, then over 60-minutes at subsequent cycles followed 60 minutes later with irinotecan 180 mg/m^2 intravenous infusion over 30 - 90 minutes. Cetuximab and Irinotecan are administered on Day 1 and Day 15 of each 28 day cycle.
Period: Overall Study
Arm/Group | Phase 1: ARQ 197+Cetuximab+Irinotecan | Phase 2: Placebo+Cetuximab+Irinotecan | Phase 2: ARQ 197+Cetuximab+Irinotecan
Started | 9 | 60 | 62
Did Not Receive Treatment | 0 | 1 | 0
Completed | 0 | 0 | 0
Not Completed | 9 | 60 | 62
Not completed — Death | 4 | 17 | 12
Not completed — Start of other or new therapy | 4 | 36 | 46
Not completed — Withdrawal by Subject | 1 | 6 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: ARQ 197+Cetuximab+Irinotecan | Phase 2: Placebo+Cetuximab+Irinotecan | Phase 2: ARQ 197+Cetuximab+Irinotecan | Total
Number analyzed (Participants) | 9 | 59 | 62 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 40 | 44 | 90
  >=65 years | 3 | 19 | 18 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (14.69) | 56.7 (12.47) | 57.4 (12.57) | 57.2 (12.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 27 | 36 | 65
  Male | 7 | 32 | 26 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 9 | 56 | 59 | 124
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Following Treatment With Tivantinib (ARQ 197) in Combination With Irinotecan and Cetuximab in Participants With Metastatic Colorectal Cancer With Wild-Type K-ras Oncogene (KRAS) Who Have Received Front-Line Systemic Therapy
Description: Progression-free survival is defined as the time from randomization to the date of disease progression (PD) or death due to any cause (as of data cutoff 12 Oct 2012).
Time Frame: Baseline up to 80 weeks postdose
Population: PFS was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Placebo+Cetuximab+Irinotecan | Phase 2: ARQ 197+Cetuximab+Irinotecan
Number analyzed (Participants) | 57 | 60
months | 7.3 [5.3 to 9.0] | 8.3 [5.6 to 10.8]
Statistical Analysis 1: Comparison: Phase 2: Placebo+Cetuximab+Irinotecan vs Phase 2: ARQ 197+Cetuximab+Irinotecan; Test type: Superiority; p = 0.3815, Log Rank
Statistical Analysis 2: Comparison: Phase 2: Placebo+Cetuximab+Irinotecan vs Phase 2: ARQ 197+Cetuximab+Irinotecan; Test type: Superiority; p = 0.1900, Peto-Peto-Prentice
Statistical Analysis 3: Comparison: Phase 2: Placebo+Cetuximab+Irinotecan vs Phase 2: ARQ 197+Cetuximab+Irinotecan; Test type: Superiority; p = 0.1986, Generalized Wilcoxon
Statistical Analysis 4: Comparison: Phase 2: Placebo+Cetuximab+Irinotecan vs Phase 2: ARQ 197+Cetuximab+Irinotecan; Test type: Superiority; p = 0.2617, Tarone-Ware

2. Primary Outcome: Progression-Free Survival (PFS) Using Computed Best Response Following Treatment With Tivantinib (ARQ 197) in Combination With Irinotecan and Cetuximab in Participants With Metastatic Colorectal Cancer Who Have Received Front-Line Systemic Therapy
Description: as for outcome 1
Time Frame: Baseline up to 80 weeks postdose
Population: PFS was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Placebo+Cetuximab+Irinotecan | Phase 2: ARQ 197+Cetuximab+Irinotecan
Number analyzed (Participants) | 57 | 60
months | 7.3 [5.3 to 9.0] | 8.3 [5.6 to 10.8]
Statistical Analysis 1: Comparison: Phase 2: Placebo+Cetuximab+Irinotecan vs Phase 2: ARQ 197+Cetuximab+Irinotecan; Test type: Superiority; p = 0.4488, Log Rank
Statistical Analysis 2: Comparison: Phase 2: Placebo+Cetuximab+Irinotecan vs Phase 2: ARQ 197+Cetuximab+Irinotecan; Test type: Superiority; p = 0.2887, Peto-Peto-Prentice
Statistical Analysis 3: Comparison: Phase 2: Placebo+Cetuximab+Irinotecan vs Phase 2: ARQ 197+Cetuximab+Irinotecan; Test type: Superiority; p = 0.1851, Generalized Wilcoxon
Statistical Analysis 4: Comparison: Phase 2: Placebo+Cetuximab+Irinotecan vs Phase 2: ARQ 197+Cetuximab+Irinotecan; Test type: Superiority; p = 0.2495, Tarone-Ware

3. Secondary Outcome: Best Overall Tumor Response and Objective Response Rate Following Treatment With Tivantinib (ARQ 197) in Combination With Irinotecan and Cetuximab in Subjects With Metastatic Colorectal Cancer Who Have Received Front-Line Systemic Therapy
Description: Best overall tumor response according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria included complete response (CR) defined as the disappearance of all target lesions; partial response (PR) defined as a ≥30% decrease in the longest diameter of target lesions; stable disease (SD) defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions. Objective response was defined as CR+PR.
Time Frame: Baseline up to 2 years 10 months postdose
Population: Best overall response and objective response rate was assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo+Cetuximab+Irinotecan | Phase 2: ARQ 197+Cetuximab+Irinotecan
Number analyzed (Participants) | 57 | 60
Participants
  Complete response (CR) | 0 | 0
  Partial response (PR) | 19 | 27
  Stable disease (SD) | 22 | 22
  Progressive disease (PD) | 13 | 9
  Objective response (CR+PR) | 19 | 27
  Inevaluable | 3 | 2

4. Secondary Outcome: Overall Survival (OS) Following Treatment With Tivantinib (ARQ 197) in Combination With Irinotecan and Cetuximab in Participants With Metastatic Colorectal Cancer With Wild-Type K-ras Oncogene (KRAS) Who Have Received Front-Line Systemic Therapy
Description: Overall survival is defined as the time from randomization date to the date of death.
Time Frame: Baseline up to 5 years 1 month postdose
Population: Overall survival was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Placebo+Cetuximab+Irinotecan | Phase 2: ARQ 197+Cetuximab+Irinotecan
Number analyzed (Participants) | 57 | 60
months
  Overall survival (12 Oct 2012 data cutoff) | 17.6 [11.3 to 20.4] | NA [13.2 to NA] — Median OS was not reached.
  Overall survival (29 Mar 2013 data cutoff) | 16.9 [12.2 to 20.4] | 19.8 [13.4 to 27.0]
  Overall survival (25 Jul 2013 data cutoff) | 16.3 [11.6 to 20.4] | 19.8 [15.4 to 27.4]
  Overall survival (20 Feb 2015 data cutoff) | 16.3 [11.6 to 20.4] | 22.3 [15.4 to 27]
Statistical Analysis 1: Comparison: Phase 2: Placebo+Cetuximab+Irinotecan vs Phase 2: ARQ 197+Cetuximab+Irinotecan; OS data cutoff as of 12 Oct 2012; Test type: Superiority; p = 0.2804, Log Rank
Statistical Analysis 2: Comparison: Phase 2: Placebo+Cetuximab+Irinotecan vs Phase 2: ARQ 197+Cetuximab+Irinotecan; OS data cutoff as of 29 Mar 2013; Test type: Superiority; p = 0.2469, Log Rank
Statistical Analysis 3: Comparison: Phase 2: Placebo+Cetuximab+Irinotecan vs Phase 2: ARQ 197+Cetuximab+Irinotecan; OS data cutoff as of 25 Jul 2013; Test type: Superiority; p = 0.1334, Log Rank
Statistical Analysis 4: Comparison: Phase 2: Placebo+Cetuximab+Irinotecan vs Phase 2: ARQ 197+Cetuximab+Irinotecan; OS data cutoff as of 20 Feb 2015; Test type: Superiority; p = 0.2159, Log Rank

5. Secondary Outcome: Duration of Response and Stable Disease Following Treatment With Tivantinib (ARQ 197) in Combination With Irinotecan and Cetuximab in Participants With Metastatic Colorectal Cancer With Wild-Type KRAS Who Have Received Front-Line Systemic Therapy
Description: Duration of response was defined for participants with complete response (CR)/partial response (PR) as the time from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of progressive disease. Duration of stable disease (SD) was defined for participants whose best response was SD at the time from the randomization date to the date of the first documentation of progressive disease. Based on Response Evaluation Criteria in Solid Tumors version 1.1, CR is defined as a disappearance of all target lesions, PR is defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Baseline up to 80 weeks postdose
Population: Duration of response and stable disease was assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Phase 2: Placebo+Cetuximab+Irinotecan | Phase 2: ARQ 197+Cetuximab+Irinotecan
Number analyzed (Participants) | 57 | 60
weeks
  Duration of response: number analyzed (Participants) | 19 | 27
  Duration of response | 29.42 (15.16) | 28.84 (16.03)
  Duration of stable disease: number analyzed (Participants) | 22 | 22
  Duration of stable disease | 24.48 (11.48) | 29.76 (15.43)

6. Secondary Outcome: Treatment-Emergent Adverse Events Reported in ≥ 10% of Participants Following Treatment With Tivantinib (ARQ 197) in Combination With Irinotecan and Cetuximab in Subjects With Metastatic Colorectal Cancer Who Have Received Front-Line Systemic Therapy
Description: A treatment-emergent adverse event (TEAE) was defined as an AE that had an onset date on or after the first dose of study drug, cetuximab, or irinotecan up to and including 30 days after the last dose of any study drug and worsened in severity after the first dose of study drug relative to the pre-treatment state.
Time Frame: Baseline up to 30 days after last dose, up to 5 years 1 month
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- All ARQ 197: All participants who received ARQ 197 treatment.
Arm/Group | Phase 1: ARQ 197+Cetuximab+Irinotecan | Phase 2: Placebo+Cetuximab+Irinotecan | Phase 2: ARQ 197+Cetuximab+Irinotecan | All ARQ 197
Number analyzed (Participants) | 9 | 59 | 62 | 71
Participants
  Any TEAE | 9 | 59 | 62 | 71
  Blood and Lymphatic System Disorders | 4 | 28 | 23 | 27
  Anaemia | 2 | 19 | 7 | 9
  Neutropenia | 4 | 13 | 18 | 22
  Gastrointestinal Disorders | 9 | 47 | 47 | 56
  Abdominal pain | 3 | 16 | 12 | 15
  Constipation | 1 | 11 | 10 | 11
  Diarrhea | 5 | 30 | 33 | 38
  Nausea | 6 | 27 | 28 | 34
  Stomatitis | 1 | 4 | 7 | 8
  Vomiting | 4 | 18 | 22 | 26
  General Disorders & Administration Site Conditions | 9 | 33 | 41 | 50
  Asthenia | 0 | 6 | 8 | 8
  Fatigue | 7 | 21 | 26 | 33
  Metabolism and Nutrition Disorders | 3 | 20 | 23 | 26
  Decreased appetite | 2 | 7 | 11 | 13
  Dehydration | 1 | 6 | 7 | 8
  Hypomagnesaemia | 2 | 6 | 6 | 8
  Nervous System Disorders | 4 | 12 | 14 | 18
  Headache | 2 | 4 | 7 | 9
  Psychiatric Disorders | 5 | 10 | 12 | 17
  Insomnia | 1 | 4 | 7 | 8
  Respiratory, Thoracic, and Mediastinal Disorders | 5 | 20 | 17 | 22
  Cough | 4 | 6 | 7 | 11
  Skin and Subcutaneous Tissue Disorders | 9 | 49 | 58 | 67
  Alopecia | 5 | 14 | 16 | 21
  Dermatitis acneiform | 4 | 9 | 8 | 12
  Dry skin | 4 | 10 | 11 | 15
  Rash | 6 | 34 | 36 | 42
  Skin fissures | 3 | 3 | 5 | 8

7. Secondary Outcome: Treatment-Emergent Infection and Infestation Adverse Events Following Treatment With Tivantinib (ARQ 197) in Combination With Irinotecan and Cetuximab in Participants With Metastatic Colorectal Cancer Who Have Received Front-Line Systemic Therapy
Description: as for outcome 6
Time Frame: Baseline up to 30 days after last dose, up to 5 years 1 month
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: ARQ 197+Cetuximab+Irinotecan | Phase 2: Placebo+Cetuximab+Irinotecan | Phase 2: ARQ 197+Cetuximab+Irinotecan | All ARQ 197
Number analyzed (Participants) | 9 | 59 | 62 | 71
Participants
  Infections and Infestations | 6 | 24 | 31 | 37
  Abscess jaw | 0 | 1 | 0 | 0
  Abscess neck | 0 | 1 | 0 | 0
  Bronchitis | 0 | 1 | 3 | 3
  Candidiasis | 1 | 0 | 0 | 1
  Cellulitis | 1 | 1 | 2 | 3
  Cystitis | 0 | 1 | 0 | 0
  Device-related infection | 1 | 0 | 0 | 1
  Diverticulitis | 0 | 0 | 1 | 1
  Ear infection | 0 | 2 | 0 | 0
  Eye infection | 0 | 0 | 2 | 2
  Folliculitis | 0 | 0 | 1 | 1
  Fungal infection | 1 | 1 | 1 | 2
  Gastroenteritis | 0 | 0 | 1 | 1
  Herpes zoster | 0 | 1 | 1 | 1
  Herpes simplex | 0 | 1 | 0 | 0
  Hordeolum | 0 | 1 | 0 | 0
  Infection | 0 | 0 | 1 | 1
  Influenza | 0 | 2 | 1 | 1
  Kidney infection | 1 | 0 | 0 | 1
  Labyrinthitis | 0 | 0 | 1 | 1
  Laryngitis | 0 | 0 | 1 | 1
  Localised infection | 0 | 1 | 0 | 0
  Nail infection | 2 | 1 | 1 | 3
  Nasopharyngitis | 0 | 1 | 2 | 2
  Oral pustule | 0 | 0 | 1 | 1
  Paronychia | 0 | 5 | 6 | 6
  Pharyngitis | 1 | 0 | 0 | 1
  Pneumonia | 1 | 1 | 1 | 2
  Pyoderma | 0 | 2 | 1 | 1
  Rash pustular | 0 | 1 | 1 | 1
  Respiratory tract infection | 0 | 0 | 2 | 2
  Respiratory tract infection viral | 0 | 1 | 2 | 2
  Sinusitis | 0 | 0 | 2 | 2
  Skin infection | 0 | 1 | 1 | 1
  Tooth abscess | 0 | 1 | 0 | 0
  Tooth infection | 0 | 2 | 0 | 0
  Tracheitis | 0 | 1 | 0 | 0
  Tracheobronchitis | 0 | 0 | 2 | 2
  Upper respiratory tract infection | 0 | 0 | 3 | 3
  Urinary tract infection | 0 | 4 | 2 | 2
  Urosepsis | 0 | 0 | 1 | 1
  Viral infection | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAE) were collected from baseline up to 30 days after last dose, up to 5 years 1 month.
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event (AE) that emerges during treatment, having been absent at pre-treatment; or reemerges during treatment, having been present at baseline but stopped prior to treatment; or worsens in severity after starting treatment relative to the pretreatment state, when the AE is continuous.
Arm/Group | Phase 1: ARQ 197+Cetuximab+Irinotecan | Phase 2: Placebo+Cetuximab+Irinotecan | Phase 2: ARQ 197+Cetuximab+Irinotecan
All-Cause Mortality (participants affected / at risk) | 6/9 | 35/59 | 35/62
Serious Adverse Events (participants affected / at risk) | 3/9 | 17/59 | 13/62
Other Adverse Events (participants affected / at risk) | 9/9 | 59/59 | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: ARQ 197+Cetuximab+Irinotecan (N=9) | Phase 2: Placebo+Cetuximab+Irinotecan (N=59) | Phase 2: ARQ 197+Cetuximab+Irinotecan (N=62)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 4 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Pneumatosis (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1
Superior vena cava occlusion (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: ARQ 197+Cetuximab+Irinotecan (N=9) | Phase 2: Placebo+Cetuximab+Irinotecan (N=59) | Phase 2: ARQ 197+Cetuximab+Irinotecan (N=62)
Anaemia (Blood and lymphatic system disorders) | 2 | 19 | 7
Leukopenia (Blood and lymphatic system disorders) | 2 | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 4 | 13 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 5
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Conjunctival irritation (Eye disorders) | 1 | 0 | 0
Ectropion (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 16 | 12
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4 | 7
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 11 | 10
Diarrhoea (Gastrointestinal disorders) | 5 | 30 | 33
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 3
Flatulence (Gastrointestinal disorders) | 0 | 5 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 5
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 27 | 28
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 4 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 4 | 7
Vomiting (Gastrointestinal disorders) | 4 | 18 | 22
Asthenia (General disorders) | 0 | 6 | 8
Chills (General disorders) | 1 | 3 | 2
Fatigue (General disorders) | 7 | 21 | 26
Hyperthermia (General disorders) | 0 | 2 | 4
Influenza-like illness (General disorders) | 1 | 1 | 0
Infusion site oedema (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 3 | 5
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 5 | 4
Pain (General disorders) | 1 | 2 | 0
Pyrexia (General disorders) | 3 | 7 | 4
Candidiasis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 2
Device-related infection (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 1 | 1
Kidney infection (Infections and infestations) | 1 | 0 | 0
Nail infection (Infections and infestations) | 2 | 1 | 1
Paronychia (Infections and infestations) | 0 | 5 | 6
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 4 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 2
Hemoglobin decreased (Investigations) | 0 | 1 | 5
Neutrophil count decreased (Investigations) | 0 | 3 | 6
Weight decreased (Investigations) | 2 | 6 | 3
White blood cell count decreased (Investigations) | 1 | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7 | 11
Dehydration (Metabolism and nutrition disorders) | 1 | 6 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 7 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 4 | 2
Headache (Nervous system disorders) | 2 | 4 | 7
Syncope (Nervous system disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 2
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 4 | 3
Insomnia (Psychiatric disorders) | 1 | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 7
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 14 | 16
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 9 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 10 | 11
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ichthyosis acquired (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Onychalgia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 6
Rash (Skin and subcutaneous tissue disorders) | 6 | 34 | 36
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 1 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 4
Skin fissures (Skin and subcutaneous tissue disorders) | 3 | 3 | 5
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Flushing (Vascular disorders) | 1 | 1 | 2
Hot flush (Vascular disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No